CLINICAL TRIAL: NCT03359252
Title: Comparison of Headache After Coil Embolization for Unruptured Intracranial Aneurysms (Standard Versus Stent-assisted): A Prospective Cohort Study
Brief Title: Headache After Coil Embolization for Unruptured Intracranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B-1710/424-304
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2021-12

CONDITIONS: Headache; Aneurysm; Endovascular Procedures
Keywords: coil embolization; headache; stent
MeSH Terms: conditions — Headache; Aneurysm

STUDY DESIGN:
Intervention Model Description: non-stent assisted coiling of unruptured intracranial aneurysms stent assisted coiling of unruptured intracranial aneurysms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-stent assisted coiling (Active Comparator): patients treated with non-stent assisted coiling of unruptured intracranial aneurysms
  Interventions: Procedure: non-stent assisted coiling
- stent assisted coiling (Experimental): patients treated with stent assisted coiling of unruptured intracranial aneurysm
  Interventions: Procedure: stent assisted coiling

INTERVENTIONS:
Procedure: non-stent assisted coiling — non-stent assisted coiling of unruptured intracranial aneurysm
  Arms: non-stent assisted coiling
Procedure: stent assisted coiling — stent assisted coiling of unruptured intracranial aneurysm
  Arms: stent assisted coiling

SUMMARY:
Perform a prospective cohort study to compare the incidence and severity of headache between non-stent assisted coiling and stent assisted coiling of unruptured intracranial aneurysms.

DETAILED DESCRIPTION:
severity of headache - assess with visual analogue scale characteristics of headache after stent deployment or simple coiling Duration of headache after intervention

ELIGIBILITY:
Inclusion Criteria:

* patients with unruptured intracranial aneurysms
* patients over 20 years old
* patients who can communicate with each other
* patients who agreed to this study (with informed consent)

Exclusion Criteria:

* patients with recurrent aneurysms after coiling or clipping
* patients with allergic reaction to antiplatelets
* patients with high risks of hemorrhage
* patients with coagulopathy
* patients with thrombocytopenia (<100,000/mm3)
* patients with liver disease (> 100 of aspartate aminotransferase or alanine aminotransferase)
* patients with renal disease (> 2mg/dL of serum creatinine)\
* patients with uncontrolled heart failure or angina
* patients with malignant tumor
* pregnant patients
* patients with past history that may associated with headache, including subarachnoid hemorrhage, head trauma, intracerebral hemorrhage, trigeminal neuralgia, arteriovenous malformation, brain tumor)
* Patients who are determined to be disqualified by researchers

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
severity of headache after coil embolization between 2 arms | prior to intervention / immediate after procedures / postoperative days 3, 7, 14, 90 days
  check change of severity of headache after coil embolization between 2 arms

SECONDARY OUTCOMES:
Duration of headache after coiling embolization after intervention | Measure the duration of time from when a headache occurs to when it disappears, assessed up to 3 months
  check duration of headache after coil embolization
characteristics of headache after coiling embolization between 2 arms | prior to intervention / immediate after procedures / postoperative days 3, 7, 14, 90 days
  identify relationship between headache location and treated aneurysm or deployed stent

CONTACTS AND LOCATIONS:
Overall Officials: O Kwon, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wiebers DO, Whisnant JP, Huston J 3rd, Meissner I, Brown RD Jr, Piepgras DG, Forbes GS, Thielen K, Nichols D, O'Fallon WM, Peacock J, Jaeger L, Kassell NF, Kongable-Beckman GL, Torner JC; International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms: natural history, clinical outcome, and risks of surgical and endovascular treatment. Lancet. 2003 Jul 12;362(9378):103-10. doi: 10.1016/s0140-6736(03)13860-3. PMID 12867109
- [Result] Sonobe M, Yamazaki T, Yonekura M, Kikuchi H. Small unruptured intracranial aneurysm verification study: SUAVe study, Japan. Stroke. 2010 Sep;41(9):1969-77. doi: 10.1161/STROKEAHA.110.585059. Epub 2010 Jul 29. PMID 20671254
- [Result] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Result] Zhang L, Wu X, Di H, Feng T, Wang Y, Wang J, Cao X, Li B, Liu R, Yu S. Characteristics of Headache After an Intracranial Endovascular Procedure: A Prospective Observational Study. Headache. 2017 Mar;57(3):391-399. doi: 10.1111/head.13006. Epub 2016 Dec 19. PMID 27991669
- [Result] Choi KS, Lee JH, Yi HJ, Chun HJ, Lee YJ, Kim DW. Incidence and risk factors of postoperative headache after endovascular coil embolization of unruptured intracranial aneurysms. Acta Neurochir (Wien). 2014 Jul;156(7):1281-7. doi: 10.1007/s00701-014-2095-8. Epub 2014 May 7. PMID 24801821